CLINICAL TRIAL: NCT04612153
Title: Musculoskeletal Disorders of Workers in a Production and Distribution Company in Argentina: a Retrospective Study
Brief Title: Musculoskeletal Disorders of Workers in a Production and Distribution Company in Argentina
Status: Completed | Type: Observational
Sponsor: Ergosol (Industry)
Responsible Party: Principal Investigator, DIEGO MENDEZ, Principal Investigator, Ergosol
Other Study IDs: EPI01
Record Dates: First submitted 2020-10-22; First posted 2020-11-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Describe Musculoskeletal Disorders of Workers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Epidemiologic — Epidemiologic study. Observational, transverse study

SUMMARY:
Describe musculoskeletal disorders of workers in a company in Argentina regarding working areas and demographic carachteristics of the workers.

DETAILED DESCRIPTION:
We are analyzing the first consultation registration of every worker that had been attended by the physiotherapist in a clinic that is located inside the company. These records consist on demographic data and also injury related information.

ELIGIBILITY:
Inclusion Criteria:

* workers in a production and distribution company in Argentina that walks into the clinic inside the company

Exclusion Criteria:

* lack of registered information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Workers with pain
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal disorders | 21 months
  Rate of participants with musculoskeletal disorders for each demographic characteristic. The measurment tool will be a face-to-face questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Mendez, PT, Principal Investigator — Ergosol
Locations (1):
- Ergosol, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No